CLINICAL TRIAL: NCT06544746
Title: Association Between Restorative Emergence Profiles and Peri-implant Bone Loss in Different Implant Systems: A Retrospective Study With up to 7 Years of Follow up
Brief Title: Association Between Restorative Emergence Profiles and Peri-implant Bone Loss in Different Implant Systems:
Status: Completed | Type: Observational
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Other Study IDs: USJ-2023-63
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Dental Implant-Abutment Designs
Keywords: Bone loss; Emergence profile; Platform switching
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone level Implants: Marginal bone loss will be assessed according to the emergence profile in each system of implants. Standardized periapical radiograph that were captured after crown placement on implants will be compared with the new radiographs done after recalling the patient.
  Interventions: Radiation: Periapical radiographs
- Tissue Level Implants: Marginal bone loss will be assessed according to the emergence profile in each system of implants. Standardized periapical radiograph that were captured after crown placement on implants will be compared with the new radiographs done after recalling the patient.
  Interventions: Radiation: Periapical radiographs

INTERVENTIONS:
Radiation: Periapical radiographs — oral radiographs taken with the paralleling technique and film holders at 1- and 3-years post-prosthesis insertion with an X-ray apparatus equipped with a long cone and a Rinn Universal Collimator (Dentsply RINN, York, PA, USA). All radiographs were stored on a PC and analyzed with the software program DBSWIN software. Each radiograph was calibrated using the implant diameter and length as reference measures to correct any distortion before measurement. An image processing program was employed to quantify peri-implant MBL, the EA, EP.

SUMMARY:
The goal of this observational study is evaluate the association between different emergence profile angulation on marginal bone loss progression around different implant systems (bone level, tissue level and switching platform).

Does different emergence profile angulation have the same effect on peri-implant marginal bone loss? Standardized periapical radiograph that were captured after crown placement on implants will be compared with the new radiographs done after recalling the patient.

DETAILED DESCRIPTION:
The present retrospective study reported the data collected on partially edentulous patients who were restored with fixed implant supported restorations. The implants were inserted in the periodontology department at the Faculty of Dental Medicine at the Saint Joseph University of Beirut, Lebanon, from 2012 to 2019. The study protocol received approval from the Institutional Review Board at Saint Joseph University of Beirut.

Under the guidance of academic members, all surgical procedures were carried out by postgraduate students. For each implant system, the surgical procedure followed the conventional recommendations. Patients got cemented or screw-retained fixed prostheses after adequate healing time of 3 to 6 months.

Patients were urged to practice proper oral hygiene after receiving their final crown. Even though all patients are told to participate in a regular Supportive periodontal therapy program, some of them did not, they were not selected and excluded in this study Patients or implants were excluded under the following conditions: (a) insufficient clinical records; (b) patients with systemic diseases or conditions; (c) smokers; (d) irregular maintenance care; (e) patients with calculus presence on radiographs; (f) implants placed on reconstructed sites; (g) implant-assisted removable prostheses; (h) peri-implantitis diagnosis; (i) failed implants;(j) Bone loss before prothesis delivery (k) previously treated peri-implantitis cases; and (l)Bone level implants placed supracrestally; (m) lack of intra-oral radiographs taken using the paralleling technique at baseline (the first year of prosthesis insertion) and after 3 years.

Patients were called for reassessment appointments after 3-7 years. After signing the informed consent, measurements by a PCP-15(periondontal probe) probe of plaque index (FMPS) and bleeding on probing (FMBS) are indicated on the form. If the smoking status has changed, it is also mentioned.

For data analysis, the following categories were included: implant connection type (bone-level platform switching, bone-level non platform switching, or tissue level); Emergence Angle (mesial and distal, separately); Emergence Profile (mesial and distal, separately); location; history of periodontitis, abutment height. Radiographic and clinical parameters taken at the time implant placement, after prosthetic delivery, and following a minimum of 3 years follow-up visit were provided.

Single and multiple restorations were included.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone the initial phase followed by implant placement.
* Implants placed and prosthesis delivered for more than 3 years.
* Implants placed in premolar/molar region
* No reconstructive bone procedure done on the site of study
* Presence of opposing occlusion
* Non-smokers

Exclusion Criteria:

* Systemic diseases (uncontrolled diabetes, drugs that can affect bone metabolism).
* Total edentulousness.
* Inappropriate, unavailable, or distorted x-rays.
* Implants placed at a supra or infra bone level.
* Implants placed immediately after an extraction.
* Poor oral hygiene (High plaque score FMPS control record > 30%)
* Smokers
* Signs of peri-implantitis development during the first year following functional loading
* Lack or incomplete information regarding peri-implant conditions (clinical and radiographic documentation at the required study time-points)
* Surgical treatment on the study implants during the first 2 years after peri-implantitis diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with implants placed and prosthesis delivered for over 3 years. Implants in the premolar/molar region. Non-smokers. Good oral hygiene. 237 implant surfaces in 76 patients. Follow-up: 3 to 7 years. Study conducted at Saint Joseph University of Beirut.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Compare Marginal Bone Loss (MBL): | Minimum of 3 years post loading
  measured mesially and distally from the implant platform until the first coronal contact of the bone with the implant. Then the total bone loss on each implant is calculated. This is achieved on the software in millimeters.
Compare Emergence angulation assessment | Minimum of 3 years post loading
  The EA was calculated as the angle between the implant's long axis and a line tangent to the restoration. First, a line parallel to the implant's long axis was drawn at the outer collar of the implant. Then, another line tangential to the restoration from the platform was drawn. The angle of intersection was measured as the emergence angle. Measured in degree
Compare Emergence profile assessment: | Minimum of 3 years post loading
  Each EP was categorized as either concave, straight, or convex.

SECONDARY OUTCOMES:
Number of Platform switching | Minimum of 3 years post loading
  Available or not
Height of Abutments | Minimum of 3 years post loading
  Height measurement of the abutment. Measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Menassa, PHD, Study Director — Saint Joseph University Of Beirut
Locations (1):
- Saint Joseph University Of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No